CLINICAL TRIAL: NCT07208630
Title: Effect of Instrument-assisted Soft Tissue Mobilization on Functional and Cognitive Abilities in Elderly
Acronym: IASTM-AGE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Nouran Ahmed Ibrahim, Nouran A. Ibrahim, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Pending2025
Record Dates: First submitted 2025-09-28; First posted 2025-10-06 (Actual); Last update posted 2025-10-06 (Actual); Status verified 2025-09

CONDITIONS: Functional Abilities; Cognitive Abilities

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- IASTM on calf muscle bilaterally plus conventional treatment (strengthening and stretching exercise (Experimental)
  Interventions: Device: Instrument-assisted soft tissue mobilization; Behavioral: Traditional physical therapy
- control group, will receive conventional treatment (Active Comparator)
  Interventions: Behavioral: Traditional physical therapy

INTERVENTIONS:
Device: Instrument-assisted soft tissue mobilization — IASTM will be delivered using stainless-steel instruments with beveled edges, applied to the target muscle groups for approximately 20 minutes per session, two times per week, over four weeks. A licensed physical therapist trained in IASTM will perform the procedure. Lubricant will be applied to the skin, and strokes will be delivered in multiple directions with pressure adapted to patient tolerance.
  Arms: IASTM on calf muscle bilaterally plus conventional treatment (strengthening and stretching exercise
Behavioral: Traditional physical therapy — The control group will receive a traditional physical therapy program focusing on strength, balance, flexibility, and functional mobility training, combined with simple cognitive stimulation tasks. Sessions will last 30 minutes, two times per week, for four weeks, supervised by a licensed physical therapist.

SUMMARY:
PURPOSE: To determine the effect of Instrument-assisted soft tissue mobilization on functional and cognitive abilities in elderly.

BACKGROUND: There is an increased interest in health care with growth of the older population.

Instrument-Assisted Soft Tissue Mobilization (IASTM) is a manual therapy technique using specially designed tools to apply pressure and mobilize soft tissues. It has gained attention as a non-invasive intervention that can aid in improving musculoskeletal health and overall function, especially in older adults. Given the aging population and the rise in age-related functional and cognitive decline, there is a pressing need for effective strategies to enhance quality of life in this demographic.

In the elderly, musculoskeletal issues, such as reduced muscle flexibility, joint stiffness, and soft tissue restrictions, are common and can severely impact physical function. IASTM has been shown to increase tissue perfusion, reduce fascial restrictions, and improve joint mobility. These effects are critical in countering age-related declines in mobility, balance, and overall physical functionality, ultimately promoting greater independence and reducing fall risk. Improved physical function through IASTM may also influence cognitive health positively, as increased physical activity and mobility are linked to better cognitive outcomes in the elderly.

HYPOTHESES: There will be no significant effect of Instrument-assisted soft tissue mobilization on functional and cognitive abilities in elderly.

RESEARCH QUESTION: Does instrument-assisted soft tissue mobilization is effective on functional and cognitive abilities in elderly?

ELIGIBILITY:
Inclusion Criteria:

60 elderly subjects aged range from 65-75 years old will participant in the study from both genders, had cognitive abilities to understand explanations and instructions, and did not take any medication that can affect their balance.

Exclusion Criteria:

they neither had sever musculoskeletal disorders nor neurological damage related to balance (dizziness, vestibular dysfunction), nor orthostatic hypotension, nor health risk factors.

Ages: 65 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-10 (Actual); Primary Completion 2025-09-15 (Actual); Study Completion 2025-10-15 (Estimated)

PRIMARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) score | Baseline and 4 weeks (end of treatment).
  Mean change in SPPB total score (0-12; higher = better physical function) from baseline to end of intervention. The SPPB includes standing balance, 4-m gait speed, and five-times-sit-to-stand.

SECONDARY OUTCOMES:
Change in Montreal Cognitive Assessment (MoCA) score | Baseline and 4 weeks (end of treatment).
  Mean change in MoCA total score (0-30; higher = better cognition) from baseline to end of intervention and at follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of physical therapy, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No